CLINICAL TRIAL: NCT04633148
Title: Multicenter, Open-label, Adaptive Design Phase I Trial With Genetically Modified T-cells Carrying Universal Chimeric Antigen Receptors (UniCAR02-T) in Combination With PSMA Peptide Target Module (TMpPSMA) for the Treatment of Patients With Progressive Disease After Standard Systemic Therapy in Cancers With Positive PSMA Marker
Brief Title: Dose-escalating Trial With UniCAR02-T Cells and PSMA Target Module (TMpPSMA) in Patients With Progressive Disease After Standard Systemic Therapy in Cancers With Positive PSMA Marker
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Although IMP has been well tolerated, biological activity was very limited. The sponsor concluded that continued development of IMP would be unlikely to result in meaningful clinical benefit for patients with prostate cancer.
Sponsor: AvenCell Europe GmbH (Industry)
Collaborators: PHARMALOG Institut für klinische Forschung GmbH (Unknown)
Responsible Party: Sponsor
Organization: AvenCell Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UC02-PSMA-01; 2019-004211-32 (EudraCT Number)
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cyclophosphamide; fludarabine; Inosine Monophosphate

STUDY DESIGN:
Intervention Model Description: Initial dose escalation followed an adaptive design. Further dose escalation includes 2 additional TMpPSMA dose levels and follows a 3+3 design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UniCAR02-T-pPSMA (Experimental): Preconditioning (lymphodepletion) with cyclophosphamide and fludarabine, followed by combination treatment of genetically modified T-cells carrying universal chimeric antigen receptors (UniCAR02-T) with the peptide TMpPSMA.
  Interventions: Drug: Cyclophosphamide (Non-IMP); Drug: Fludarabine (Non-IMP); Drug: UniCAR02-T-pPSMA; Drug: UniCAR02-T (IMP)

INTERVENTIONS:
Drug: Cyclophosphamide (Non-IMP) — Intravenous infusion for 3 days
Drug: Fludarabine (Non-IMP) — Intravenous infusion for 3 days
Drug: UniCAR02-T-pPSMA — Intravenous Infusion for 21 days
Drug: UniCAR02-T (IMP) — Intravenous infusion of single dose

SUMMARY:
This dose-escalating phase I trial assesses for the first time the safety, the side effects and the harmlessness, as well as the therapeutical benefit of the new study drug UniCAR02-T-pPSMA in patients with progressive disease after standard systemic therapy in castration-resistant prostate cancers with positive PSMA marker. The UniCAR02-T-pPSMA drug is a combination of a cellular component (UniCAR02-T) with a recombinant antibody derivative (TMpPSMA) which together forms the active drug.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients diagnosed with progressive castration-resistant prostate cancer refractory to standard treatments and with no other available standard or curative treatment
3. Measurable or non-measurable disease based on immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) and positivity in PSMA Positron Emission Tomography (PET)
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
5. Life expectancy of at least 3 months
6. Adequate renal and hepatic laboratory assessments
7. Adequate cardiac function, i.e. left ventricular ejection fraction (LVEF)
8. Permanent venous access existing (e.g. port-system) resp. acceptance of implantation of a device
9. Able to give written informed consent
10. Weight ≥ 45kg
11. Using a highly effective method of birth control

Exclusion Criteria:

1. Central nervous system metastasis or meningeosis carcinomatosa
2. Cardiac disease: i.e. heart failure (NYHA III or IV); unstable coronary artery disease, myocardial infarction or serious cardiac ventricular arrhythmias requiring anti-arrhythmic therapy within the last 6 months prior to study entry
3. Patients undergoing renal dialysis
4. Pulmonary disease with clinical relevant hypoxia (need for oxygen inhalation)
5. Parkinson, epilepsy and stroke or presence or history of seizures, paresis, aphasia, central nervous system (CNS) or intracranial hemorrhage
6. History or presence of disseminated intravascular coagulation (DIC) or thromboembolism within the last three months
7. Multiple sclerosis
8. Hemolytic anemia
9. Eye diseases with neovascularization
10. Active infectious disease considered by investigator to be incompatible with protocol or being contraindications for lymphodepletion therapy
11. Presence of urotoxicity from previous chemo- or radiotherapy or urinary outflow obstruction
12. Vaccination with live viruses less than 2 weeks prior lymphodepletion therapy
13. Any disease requiring immunosuppressive therapy
14. Major surgery within 28 days (prior start of TMpPSMA infusion)
15. Other malignancy requiring active therapy but adjuvant endocrine therapy is allowed
16. Treatment with any investigational drug substance or experimental therapy within 4 weeks or 5 half-lives of the substance (whatever is shorter) prior to administration of TMpPSMA
17. Prior treatment with gene therapy products
18. Use of checkpoint inhibitors within 5 half-lives of the respective substance prior to administration of TMpPSMA
19. Autoimmune diseases requiring systemic steroids or other systemic immunosuppressants (note that physiologic steroid replacement not exceeding 10 mg prednisolone equivalent per day is allowed)
20. Psychologic disorders, drug and/or significant active alcohol abuse
21. Known history of human immunodeficiency virus (HIV) or active/chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV)
22. Presence of autoantibodies against La/SS-B or presence or history of autoimmune diseases (e.g. systemic lupus erythematosus, SS/SLE overlap syndrome, subacute cutaneous lupus erythematosus, neonatal lupus, primary biliary cirrhosis, Sjögren's syndrome)
23. Known hypersensitivity to cellular component (UniCAR02-T) and/or targeting peptide module (TMpPSMA) excipients and/or contraindication to compounds of the lymphodepletion therapy (cyclophosphamide and fludarabine), and tocilizumab or corticosteroids as specified in the respective IB/SmPC
24. Evidence suggesting that the patient is not likely to follow the study protocol (e.g. lacking compliance)
25. Incapability of understanding purpose and possible consequences of the trial
26. Patients who should not be included according to the opinion of the investigator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | DLT period (infusion period of TMpPSMA + 7 days or + 14 days in patients with with myelosuppression)
  Incidence and intensity of adverse events graded according to CTCAE V5.0 with the exception of CRS and ICANS graded according to Lee et al. 2014 and Lee et al. 2019 respectively
Incidence of dose limiting toxicity (DLT) | DLT period (infusion period of TMpPSMA + 7 days or + 14 days in patients with with myelosuppression)
  DLT is defined as any adverse event at least possible related to TMpPSMA and/or UniCAR02-T
Maximum tolerated dose (MTD) | DLT period (infusion period of TMpPSMA + 7 days or + 14 days in patients with with myelosuppression)
  The dose for which the isotonic estimate of the DLT probability is closest to the target DLT probability of 0.2.

SECONDARY OUTCOMES:
Recommended phase 2 dose (RP2D) | DLT period (infusion period of TMpPSMA + 7 days or + 14 days in patients with with myelosuppression)
  The RP2D will be determined based on MTD, all available efficacy data, and all available safety data, including information derived from additional treatment cycles.
Antitumor activity | DLT period (infusion period of TMpPSMA + 7 days or + 14 days in patients with with myelosuppression)
  Antitumor activity of UniCAR02-T-pPSMA at any time point according to irRECIST (immune-related) Response Evaluation Criteria in Solid Tumors): Complete remission (CR) and partial remission (PR), Objective response rate (ORR), Disease control rate (DCR), Best response rate, Duration of response (DOR),Progression free survival (PFS)
Prostate specific antigen (PSA) response | DLT period (infusion period of TMpPSMA + 7 days or + 14 days in patients with with myelosuppression)
Overall Survival (OS) | Until fifteen years after last UniCAR02-T administration
Influence on Circulating tumor cells (CTC) | Before start of lymphodepletion therapy until 6 resp. 12 months after start of last TMpPSMA application

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Bargou, Prof., Principal Investigator — Wuerzburg University Hospital
Locations (4):
- Germany (4):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No